CLINICAL TRIAL: NCT06232252
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Intravenous Doses of BI 765423 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Well Multiple Doses of BI 765423 Are Tolerated by Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1493-0008; 2023-506722-36-00 (Registry Identifier: CTIS); U1111-1298-0452 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: The groups will be dosed sequentially. Within each dose group, some subjects will receive BI 765423 and some will receive placebo.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant: This trial is blinded to treatment but not to dose level. The dose level will be known to the participant.
  Outcome assessor: ECG laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose group (DG) 1 (very low dose) (Experimental)
  Interventions: Drug: BI 765423; Drug: Placebo matching BI 765423
- Dose group (DG) 2 (low dose) (Experimental)
  Interventions: Drug: BI 765423; Drug: Placebo matching BI 765423
- Dose group (DG) 3 (medium dose) (Experimental)
  Interventions: Drug: BI 765423; Drug: Placebo matching BI 765423
- Dose group (DG) 4 (high dose) (Experimental)
  Interventions: Drug: BI 765423; Drug: Placebo matching BI 765423

INTERVENTIONS:
Drug: BI 765423 — BI 765423
Drug: Placebo matching BI 765423 — Placebo matching BI 765423

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics of BI 765423 in healthy male subjects.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), respiratory rate (RR), temperature), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body Mass Index (BMI) of 18.5 to 29.9 kg/m² (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
5. Male subjects who are willing to not donate sperm for the duration of the trial until completion of EoS visit and meet at least one of the following criteria:

   * Not sexually active with a partner of child-bearing potential or sexually abstinent. Women of non-childbearing potential are defined as postmenopausal for at least 1 year or surgically sterilised by hysterectomy, bilateral salpingectomy or bilateral oophorectomy. True abstinence is only acceptable, if it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active, but becomes active with their partner, they must comply with the contraceptive requirements detailed below.
   * Sexually active with a partner of child-bearing potential who is willing to use combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom in male subject from Screening until at least end of study (EoS) visit.
   * Sexually active with a partner of child-bearing potential who is willing to use progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom in male subject from Screening until at least EoS visit.
   * Sexually active with a partner of child-bearing potential who is willing to use intrauterine device (IUD) or intrauterine hormone-releasing system (IUS), plus condom in male subject from Screening until at least EoS visit.
   * Male subject is vasectomised (vasectomy at least 1 year prior to enrolment) and received medical assessment of the surgical success (documented absence of sperm). If sexually active with a partner of child-bearing potential, the subject is willing to use male condom from Screening until at least EoS visit.

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR, RR, temperature or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm) (subjects with heart rate values between 45 and 50 bpm may be enrolled in case they have a normal thyroid function, no clinical symptoms associated with the bradycardia and no apparent signs of other diseases causing bradycardia such as hypothyroidism)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Major surgery (major according to the investigator's assessment) performed within 3 months prior to screening or planned after screening during the study, e.g. hip replacement
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects treated with BI 765423 who experience any treatment-emergent adverse event assessed as drug-related by the investigator | up to 145 days for DG 1 and 2, up to 159 days for DG 3 and 4

SECONDARY OUTCOMES:
AUCτ (area under the concentration-time curve of the analyte in serum over a uniform dosing interval τ) | up to 336 hours for DG 1 and 2, up to 673 hours for DG 3 and 4
Cmax (maximum measured concentration of the analyte in serum) | up to 141 days for DG 1 and 2, up to 155 days for DG 3 and 4

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com